CLINICAL TRIAL: NCT01741636
Title: Survivorship Care Planning in Colorectal and Lung Cancer: A Feasibility Study
Brief Title: Survivorship Care Planning in Patients With Colorectal or Non-Small Cell Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 12342; NCI-2012-02783 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-12-03; First posted 2012-12-05 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2013-12

CONDITIONS: Stage I Colon Cancer; Stage I Rectal Cancer; Stage IA Non-small Cell Lung Cancer; Stage IB Non-small Cell Lung Cancer; Stage IIA Colon Cancer; Stage IIA Non-small Cell Lung Cancer; Stage IIA Rectal Cancer; Stage IIB Colon Cancer; Stage IIB Non-small Cell Lung Cancer; Stage IIB Rectal Cancer; Stage IIC Colon Cancer; Stage IIC Rectal Cancer; Stage IIIA Colon Cancer; Stage IIIA Non-small Cell Lung Cancer; Stage IIIA Rectal Cancer; Stage IIIB Colon Cancer; Stage IIIB Non-small Cell Lung Cancer; Stage IIIB Rectal Cancer; Stage IIIC Colon Cancer; Stage IIIC Rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Early Intervention, Educational; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Supportive care (survivorship plan) (Experimental): Patients undergo Survivorship Care Planning comprising disease surveillance, management of potential long-term and late effects, psycho-social-spiritual issues, and healthy living recommendations.
  Interventions: Other: educational intervention; Other: questionnaire administration; Procedure: quality-of-life assessment

INTERVENTIONS:
Other: educational intervention — Undergo Survivorship Care Planning
  Other Names: intervention, educational
Other: questionnaire administration — Ancillary studies
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment

SUMMARY:
Survivorship Care Planning may improve overall well-being and quality of life of colorectal and lung cancer survivors

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To test the feasibility and acceptability of an Advanced Practice Nurse (APN) driven Survivorship Care Planning (SCP) intervention for colorectal cancer (CRC) and non-small cell lung cancer (NSCLC) survivors.

SECONDARY OBJECTIVES:

I. Development of the infrastructure and strategy for a larger comparative intervention study.

OUTLINE:

Patients undergo Survivorship Care Planning comprising disease surveillance, management of potential long-term and late effects, psycho-social-spiritual issues, and healthy living recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed diagnosis of stage I, II, or III CRC or NSCLC
* Able to read and understand English
* Able to read and/or understand the study protocol requirements, and provide written informed consent
* Diagnosis of CRC or NSCLC
* Within three months of completing primary treatment (surgery, chemotherapy, radiation, or chemoradiation)
* Without recurrent or new primary cancers

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Percentage of attrition based on number of patients who failed to complete the two-month study | 2 months
  Descriptive statistics will be presented on those who agree to participate and the proportion of those approached who agree to participate.
Total retention across the two month follow-up | 2 months
  Descriptive statistics will be presented on those who agree to participate and the proportion of those approached who agree to participate.
Percentage of those who are qualified and agree to participate | 2 months
Data collection protocols including who will administer the survey, timing of surveys, telephone interviews vs. face to face administration | 2 months
Cost implications including hiring and training of the research staff, development of study manuals and patient education materials, research staff time, intervention supplies, and other miscellaneous costs | 2 months
Satisfaction with the timing, content, and delivery of the intervention | 2 months
  Quantitative and qualitative descriptive statistics will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Sun, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States